CLINICAL TRIAL: NCT03929952
Title: Descriptive Pilot Study of the Effects of a Standardized Neuromodulation Program on Cortical Brain Function in Chronic Low Back Pain Patients
Acronym: NEMOLOC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: NIMAO/2018-01/AD-01; 2021-A00437-34 (Other: ANSM)
Record Dates: First submitted 2019-04-24; First posted 2019-04-29 (Actual); Last update posted 2025-01-07 (Actual); Status verified 2025-01

CONDITIONS: Low Back Pain; Chronic Low Back Pain
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Chronic low back pain (Experimental)
  Interventions: Other: Neurofeedback treatment; Other: functional magnetic resonance imaging (fMRI) scans

INTERVENTIONS:
Other: Neurofeedback treatment — 20 sessions of neurofeedback of 5 minutes each consisting of :
  * The patient is equipped with an electroencephalography headset. The feedback visual has the form of a candle flame and is modulated by alpha synchrony.
  * The height of the flame is proportional to the intensity of the patient's pain. The patient has to concentrate on the height of this flame by thought to modulate it and, at the same time, to decrease the intensity of his own pain.
Other: functional magnetic resonance imaging (fMRI) scans — The patient in alpha synchrony related state and in rating state will undergo an fMRI

SUMMARY:
This study aims to evaluate neurofeedback-induced changes in brain function and the correlations between these changes and clinical scores by functional magnetic resonance imaging and electroencephalography in patients with low back pain.

ELIGIBILITY:
Inclusion Criteria:

* Patient with a wifi connexion at home
* Patient with the ability to modulate the height of the candle by thinking in the alpha synchrony test.
* Patient with chronic low back pain for more than six months with a visual analogue pain scale greater than 5 impacting activities of daily living, hobbies and work
* Patient having given free and informed consent and signed consent.
* Affected patient or beneficiary of a health insurance plan.
* Patient who is at least 18 years old (≥) and younger than 75 years old (<).

Exclusion Criteria:

* Pregnant or breastfeeding patient
* Patient with a contraindication to performing a fMRI scan: ferromagnetic implant in the body, piercing, claustrophobia, unable to remain in the scanner stationary for 40 minutes
* Patient already included in another study
* Patient in a exclusion period determined by a previous study
* The subject is under the protection of justice, guardianship or curatorship.
* The subject refuses to sign the consent.
* It is not possible to give the subject informed information.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2022-01-19 (Actual); Primary Completion 2024-10-25 (Actual); Study Completion 2024-10-25 (Actual)

PRIMARY OUTCOMES:
Description of the cortical zone activated by neurofeedback | Day 20
  Measure taken by electroencephalography

SECONDARY OUTCOMES:
Back Beliefs Questionnaire (BBQ) | Day 20
  Auto-Questionnaire with 14 items describing the patient beliefs about chronic low back pain. The higher the score, the more the beliefs are negative
Fear Avoidance Beliefs Questionnaire (FABQ) | Day 20
  Auto-Questionnaire with 16 items describing apprehension and avoidance in relation to professional activities and physical activities.
Oswestry Disability Index (ODI) | Day 20
  Scale used to assess the functional disability of low back pain patients.
Coping Strategies Questionnaire (CSQ) | Day 20
  Auto-Questionnaire with 21 items evaluating coping strategies specific to pain and especially in low back pain
Hospital Anxiety and Depression Scale (HADS) | Day 20
  Auto-Questionnaire with 14 items used in the detection of anxio-depressive disorders. The higher the score, the more the depression is severe.
Scale of lumbar pain in Quebec | Day 20
  Autoquestionnaire with 20 items used to measure the functional repercussions of low back pain on simple actions of everyday life. The higher the score, the more low back pains have a significant functional impact.
Tampa scale | Day 20
  Autoquestionnaire with 17 items used to estimate the level of kinesiophobia (fear and fear) related to pain that leads to avoidance of activities considered to cause or increase pain or to cause or aggravate an injury. The higher the score, the higher the level of kinesiophobia.

CONTACTS AND LOCATIONS:
Overall Officials: Arnaud Dupeyron, MD, Principal Investigator — Nîmes University Hospital
Locations (1):
- Nimes University Hospital, Nîmes, France